CLINICAL TRIAL: NCT03708276
Title: Testing a New Multiple Sclerosis Specific Web-based Symptom Self-management Program: My MS Toolkit
Brief Title: My MS Toolkit: a Symptom Self-management Program for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anna Kratz, Associate Professor of Physical Medicine and Rehabilitation, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00146844; W81XWH-17-1-0367 (Other: United States Department of Defense)
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: Self-management; Web-based program
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My MS Toolkit (Experimental): 20 Participants asked to use My MS Toolkit.
  Interventions: Other: My MS Toolkit

INTERVENTIONS:
Other: My MS Toolkit — My MS Toolkit, a web-based self-management intervention designed to help persons with Multiple Sclerosis self-manage fatigue, pain, and depressed mood.

SUMMARY:
My MS Toolkit is a web-based symptom self-management program for persons with multiple sclerosis.

This study is evaluating various aspects of My MS Toolkit and how it impacts symptom self-management in multiple sclerosis. The research team believe that the toolkit will be feasible, acceptable, and beneficial to participants.

DETAILED DESCRIPTION:
Study participants will be asked to use a newly developed web-based symptom self-management program, called the My MS Toolkit, for 12 weeks. Participants will also be asked to complete online surveys throughout the study.

The My MS Toolkit includes 8 modules that describe symptom self-management strategies. Participants will explore the My MS Toolkit on their own, following the prompts and guides built into the program, and are encouraged to practice and apply the skills learned.

The study can be done from participants' homes using a reliable internet-connected device. No travel is required.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* Have access to a reliable, internet-connected device (e.g. computer, tablet). (Note: this study is conducted electronically and is not location dependent.)
* One or more of the following:

  1. Moderate/moderately severe depressive symptoms
  2. Chronic pain
  3. Presence of significant fatigue symptoms
* Read, speak and understand English.

Exclusion Criteria:

* Significant cognitive impairment
* Current psychotherapy for symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Acceptability of My MS Toolkit | week 12-week 14
  Assessed by the Patient Satisfaction Evaluation Scale, 12 question scale where each response score ranges from 4 to 1 and the total score ranges from 48 to 12. Higher scores indicate increased satisfaction.
Feasibility of My MS Toolkit | up to week 12
  Assessed by the treatment adherence questionnaire that consists of 5 questions that assess: 1) how many times the participant accessed the website in the prior two weeks; 2) how many minutes the participant spent on the website; 3) which parts of the website the participant accessed; 4) which activities the participant engaged in; and 5) which skill from the website the participant used. The items on this questionnaire will be used to describe the use of the website for assessing treatment adherence by participants in the study.

SECONDARY OUTCOMES:
Impact of My MS Toolkit: Change in fatigue | Pre- and post-treatment, up to 14 weeks
  The Modified Fatigue Impact Scale will be used to assess fatigue. It is a self-report survey that contains 21 items. Each item is rated 0-4. Higher scores indicate a greater impact of fatigue on a person's activities.
Impact My MS Toolkit: Change in pain interference | up to 14 weeks
  The BPI-SF is a 9-item questionnaire (15 prompts) with two domains: pain severity and pain interference. The 7 pain interference items have values which range from 0 ("does not interfere") to 10 ("completely interferes"); items are averaged for a scale score range of 0-10, with higher scores indicating more pain interference.
Impact My MS Toolkit: Change in depressive symptoms | up to 14 weeks
  The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. Scores range from 0 - 24 and a score of 10 or greater is consistent with at least moderate depressive symptoms.
Change in self-efficacy for managing symptoms | up to 14 weeks
  Changes measured by the University of Washington Self-Efficacy Scale (UW-SES), higher score indicates higher levels of self-efficacy (total score range: 6-30)
Participant perception of change | week 12-14
  Perception of change is assessed by the patient global impression of change questionnaire, which is 1 question and responses range from 1-7. Higher numbers indicate greater improvement in condition.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kratz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kratz AL, Alschuler KN, Williams DA, Ehde DM. Development and pilot testing of a web-based symptom management program for multiple sclerosis: My MS toolkit. Rehabil Psychol. 2021 May;66(2):224-232. doi: 10.1037/rep0000375. Epub 2021 Feb 4. PMID 33539138

DOCUMENTS (1):
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03708276/ICF_000.pdf